CLINICAL TRIAL: NCT05103124
Title: Efficacy of GUM Hydral Mouthwashes on Symptoms of Radiotherapy-induced Xerostomia: a Randomized, Double-blind, Crossover Study.
Brief Title: GUM Hydral Mouthwash vs Placebo in the Management of Hyposalivation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Sunstar Italiana SRL. (Unknown)
Responsible Party: Principal Investigator, Carlo Lajolo, Associate Professor and Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SSHNC-1
Record Dates: First submitted 2021-10-17; First posted 2021-11-02 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Xerostomia; Xerostomia Following Radiotherapy
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydral (Experimental): The participants will be asked to rinse their mouth five times a day with the experimental product. After one month, the administration will be stopped and the patients will be asked to fulfill the questionnaires mentioned in the methods section (XQ, QLQ-C30, QLQ HN35)
  Interventions: Device: Hydral; Other: Placebo
- Placebo (Placebo Comparator): The participants will be asked to rinse their mouth five times a day with the placebo comparator. After one month, the administration will be stopped and the patients will be asked to fulfill the questionnaires mentioned in the methods section (XQ, QLQ-C30, QLQ HN35)
  Interventions: Device: Hydral; Other: Placebo

INTERVENTIONS:
Device: Hydral — The investigational product GUM Hydral will be administered for a 30-days treatment period
Other: Placebo — The placebo product will be administered for a 30-days treatment period

SUMMARY:
There is currently little robust evidence to inform the management of hyposalivation and xerostomia in this population. Although the treatment of xerostomia is very individual, a first-line medication is needed to ameliorate the dehydration in the mouth by substituting for the secretion of saliva.

The aim of this study is to describe the effect of the administration of Hydral on reducing patients' xerostomia symptoms due to radiotherapy.

The study will be conducted as a double-blind randomized clinical trial (RCT) and foresees a crossover design, so the population will be divided into two groups, receiving both the medical device and the placebo.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) accounts for more than 750,000 new cases per year and its prognosis is still poor in terms of mortality and of morbidity and it causes approximately 350,000 deaths annually worldwide. Radiotherapy (RT) is an established treatment modality for HNSCC and other H&N tumors, either for treatment alone or as adjuvant. Unfortunately, high-dose RT has significant adverse effects on the oral and maxillofacial tissues, both hard and soft. In particular, when salivary glands are within the irradiated field, irreversible salivary glands damage occurs in 63-93% of the patients. Salivary gland damage typically manifests as reduced saliva secretion, which in turn can translate into a subjective sensation of dry mouth (xerostomia), oral discomfort, altered taste, difficulty with speaking, swallowing, chewing, and increased risk of dental disease. Overall hyposalivation and related xerostomia can cause a substantial reduction in quality-of-life (QoL). However there is currently little robust evidence to inform the management of hyposalivation and xerostomia in this population. Although the treatment of xerostomia is very individual, a first-line medication is needed to ameliorate the dehydration in the mouth by substituting for the secretion of saliva.

GUM Hydral (GUM Hydral: Sunstar Italiana SRL. Corso Italia 13 21047 Saronno, VA, Italy) is a product based on hyaluronic acid and sodium citrate. It helps in rehydrating and protecting the oral tissues, by forming a film on those tissues. It may be helpful in reducing the xerostomia symptoms.

The device is a high-density liquid and it is used as a mouthwash. In this trial, the aim is to investigate if its efficacy in reducing the xerostomia symptoms is higher than placebo.

The placebo will be made of water with xylitol in addition. Xylitol is a is a sugar alcohol used as a sugar substitute, which does not increase the risk of tooth decay. In this formulation, its only role is to give a slight sweet flavor to water.

The aim of this study is to describe the effect of the administration of Hydral on reducing patients' xerostomia symptoms due to radiotherapy.

The study will be conducted as a double-blind randomized clinical trial (RCT) and foresees a crossover design, so the population will be divided into two groups, receiving both the medical device and the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the informed consent form
* Patients older than 18 years
* Patients with diagnosis of HNC, who had received local radiotherapy at least three months before the beginning of the study, involving the salivary glands, both for curative and palliative purpose, with or without chemotherapic treatment, reporting xerostomia symptoms
* Patients with diagnosis of HNC, who had received local radiotherapy as an adjuvant to surgical resection at least three months before the beginning of the study, with or without chemotherapic treatment, reporting xerostomia symptoms-

Exclusion Criteria:

* Patients with documented contraindication to any of the components of GUM HYDRAL (there included eccipients)
* Patients with any neurological and psychiatric condition having an influence on the ability to self-apply the treatment
* Patients unwilling to complete the request diary card
* Patients unable to attend the ambulatory visits scheduled by the protocol
* Patients participating to other clinical studies
* Patients who had received antitumoral treatment during the previous three months
* Patients with concomitant Sjogren's syndrome
* Other causes of xerostomia (pharmacological treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Improvement of the Xerostomia Questionnaire (XQ) | After a one-month therapy both with Hydral and Placebo
  The modified XQ provides a measure of the severity of radiation -induced xerostomia that affects the patients' QoL. This questionnaire consists of 10 questions, associated with patient-reported dryness. Moreover, a general question "how dry is your mouth?" has been added to the questionnaire. The modified XQ is a self-administered tool and patients will be asked to rate each symptom on a 10-point NRS scale of 0-10, with higher scores indicating more severe dryness or discomfort due to dryness. Each item score is added, and the sum is linearly transformed to produce the final summary score ranging from 0 to 100, with higher scores representing higher levels of xerostomia.

SECONDARY OUTCOMES:
Improvement of the EORTC QLQ-30 questionnaire | After a one-month therapy both with Hydral and Placebo
  The QLQ-C30 provides 30 questions, globally assessing patients' quality of life. The answers will be converted into a linear scoring scale, with values between 0 and 100, as advocated by EORTC.
Improvement of the EORTC QLQ_H&N-35 Questionnaire | After a one-month therapy both with Hydral and Placebo
  The QLQ-H&N35 includes 35 questions, and addresses symptoms associated with specific tumor location, side effects associated with the oncologic treatment and additional QoL aspects modified by the disease or its treatment. The answers will be converted into a linear scoring scale, with values between 0 and 100, as advocated by EORTC.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lajolo, Prof., Principal Investigator — CU Sacred Hearth
Locations (1):
- Catholic University of the Sacred Hearth, Roma, Italy

REFERENCES:
- [Derived] Rupe C, Basco A, Gioco G, Patini R, Lucchese A, Micciche F, Massaccesi M, Lajolo C. Sodium-hyaluronate mouthwash on radiotherapy-induced xerostomia: a randomised clinical trial. Support Care Cancer. 2023 Oct 18;31(12):644. doi: 10.1007/s00520-023-08090-x. PMID 37851095

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT05103124/Prot_SAP_000.pdf